CLINICAL TRIAL: NCT02291250
Title: Effect of Soft Fruit on Postprandial Blood Glucose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Rowett 905
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
Keywords: anthocyanin; blackcurrant; greencurrant; glucose; polyphenol; post prandial glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sugar matched water with polycal OGTT (Experimental): 1. Control: sugar matched (matched to currant sugar content) water with polycal
  2. Blackcurrants (200grams) with polycal
  3. Blackcurrants (200grams) with glucose
  4. Greencurrants (200grams) with polycal Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The OGTT will be carried out with glucose as a simple carbohydrate load or polycal as a complex carbohydrate load.
  Volunteers will be randomised into four groups (n=4 per group). One week wash out between treatments
  Interventions: Dietary Supplement: Sugar matched water with polycal OGTT
- Blackcurrants with polycal OGTT (Experimental): 1. Blackcurrants (200grams) with polycal
  2. Blackcurrants (200grams) with glucose
  3. Greencurrants ( 200grams) with polycal
  4. Control: sugar matched (matched to currant sugar content) water with polycal
  Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The OGTT will be carried out with glucose as a simple carbohydrate load or polycal as a complex carbohydrate load as decribed above.
  Volunteers will be randomised into four groups (n=4 per group). One week wash out between treatments
  Interventions: Dietary Supplement: Blackcurrants with polycal OGTT
- Blackcurrants with glucose OGTT (Experimental): 1. Blackcurrants (200grams) with glucose
  2. Greencurrants (200grams) with polycal
  3. Control: sugar matched (matched to currant sugar content) water with polycal
  4. Blackcurrants (200grams) with polycal
  Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The OGTT will be carried out with glucose as a simple carbohydrate load or polycal as a complex carbohydrate load as decribed above
  Volunteers will be randomised into four groups (n=4 per group). One week wash out between treatments
  Interventions: Dietary Supplement: Blackcurrants with glucose OGTT
- Greencurrants with polycal OGTT (Experimental): 1. Greencurrants (200grams) with polycal
  2. Control: sugar matched (matched to currant sugar content) water with polycal
  3. Blackcurrants (200grams) with polycal
  4. Blackcurrants (200grams) with glucose
  Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The OGTT will be carried out with glucose as a simple carbohydrate load or polycal as a complex carbohydrate load as decribed above.
  Volunteers will be randomised into four groups (n=4 per group). One week wash out between treatments.
  Interventions: Dietary Supplement: Greencurrants with polycal OGTT

INTERVENTIONS:
Dietary Supplement: Blackcurrants with polycal OGTT — Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The consumption of the currants will be followed by an oral glucose tolerance test (OGTT) with Polycal (complex carbohydrate) or glucose (simple carbohydrate) as the carbohydrate load.
  The equivalent carbohydrate load will be standardised across the groups
  Arms: Blackcurrants with polycal OGTT
Dietary Supplement: Greencurrants with polycal OGTT — Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The consumption of the currants will be followed by an oral glucose tolerance test (OGTT) with Polycal (complex carbohydrate) or glucose (simple carbohydrate) as the carbohydrate load.
  The equivalent carbohydrate load will be standardised across the groups
  Arms: Greencurrants with polycal OGTT
Dietary Supplement: Blackcurrants with glucose OGTT — Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The consumption of the currants will be followed by an oral glucose tolerance test (OGTT) with Polycal (complex carbohydrate) or glucose (simple carbohydrate) as the carbohydrate load.
  The equivalent carbohydrate load will be standardised across the groups
  Arms: Blackcurrants with glucose OGTT
Dietary Supplement: Sugar matched water with polycal OGTT — Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.
  The consumption of the currants will be followed by an oral glucose tolerance test (OGTT) with Polycal (complex carbohydrate) or glucose (simple carbohydrate) as the carbohydrate load.
  The equivalent carbohydrate load will be standardised across the groups
  Arms: Sugar matched water with polycal OGTT

SUMMARY:
Dietary strategies for alleviating health complications associated with type 2 diabetes (T2D) are being pursued as alternatives to pharmaceutical interventions. Berries such as blackcurrants that are rich in polyphenols may influence carbohydrate digestion and absorption and thus postprandial glycaemia. In addition berries have been reported to alter incretins as well as to have anti-oxidant and anti-inflammatory properties that may also affect postprandial glycaemia. This study investigated the acute affect blackcurrants on glucose metabolism in overweight/obese volunteers .

DETAILED DESCRIPTION:
Sixteen overweight/obese volunteers from the Aberdeen area will be recruited into a randomised controlled study. Volunteers will be randomised into four groups matched for BMI and age and given 200 grams of blackcurrants (which contain anthocyanins) or greencurrants (which naturally contain no anthocyanins), followed by an OGTT.

The consumption of the currants will be followed by an oral glucose tolerance test (OGTT) with Polycal (complex carbohydrate) or glucose (simple carbohydrate) as the carbohydrate load.

There will be a one week minimum wash out period between each intervention. All interventions will be randomised and blinded as far as possible in a cross-over design where the volunteers are acting as their own control. The volunteers will be asked to consume a low phytochemical diet three days prior to taking the currants all occasions. In addition, they will be asked to record what they ate over the same period in a simple food diary.

The following intervention will be carried out on 16 overweight/obese male/postmenopausal female non-smoker volunteers:

1. Control: sugar matched (matched to currant sugar content) water with polycal (complex carbohydrate load)
2. Blackcurrants (which contain anthocyanins; 200grams) with polycal (complex carbohydrate load)
3. Blackcurrants (which contain anthocyanins; 200grams) with glucose (simple carbohydrate load)
4. Greencurrants (which naturally contain no anthocyanins; 200grams) with polycal (complex carbohydrate load)

Note: the polycal will contain the equivalent glucose load as given in intervention 3 assuming complete hydrolysis of all carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* Obese male or female (postmenopausal) healthy non-smoking volunteers (BMI over 25kg/m2)
* Aged >21 and <70 years

Exclusion Criteria:

* Medical exclusion criteria
* Chronic illness, including:

  * thromboembolic or coagulation disease
  * unregulated thyroid disease
  * kidney disease
  * hepatic disease
  * severe gastrointestinal disorders
  * pulmonary disease (e.g. chronic bronchitis, COPD)
  * diabetes
* Alcohol or any other substance abuse
* Eating disorders
* Psychiatric disorders (including severe depression, lithium treatment, schizophrenia, severe behavioural disorders)
* Non-postmenopausal women
* Medication exclusion criteria
* Oral steroids
* Tricyclic antidepressants, neuroleptics
* Anticoagulants
* Digoxin and anti-arrhythmics
* Chronic use of anti-inflammatories (e.g. high doses of aspirin, ibuprofen), Insulin, -Sulphonylureas, Thiazolidinediones (glitazones), metformin.
* Anti-obesity medication e.g. Orlistat

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-11; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Plasma Glucose Area Under the Curve | Plasma was collected at -15, -10 and -5 (fasted) and at 15, 30, 45, 60, 90, 120, 150 and 300 min post currant ingestion

SECONDARY OUTCOMES:
Plasma Insulin Area Under the Curve | Plasma was collected at -15, -10 and -5 (fasted) and at 15, 30, 45, 60, 90, 120, 150 and 300 min post currant ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided